CLINICAL TRIAL: NCT05157087
Title: XOLAIR (Omalizumab) Outcomes in Pediatric Allergic Asthma Patients in the United States
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CIGE025AUS55
Record Dates: First submitted 2021-11-30; First posted 2021-12-14 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Asthma
Keywords: Asthma,; Omalizumab (Xolair),; Asthma Control,; Corticosteroids,; Pediatric,; Children,; Adolescents,; Healthcare Expenditures
MeSH Terms: conditions — Asthma | interventions — Omalizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Commercial Population: Individuals with at least one omalizumab prescription in the Marketscan commercial claims during the identification period (07/07/2016 - 12/31/2018)
  Interventions: Drug: Omalizumab
- Medicaid Population: Individuals with at least one omalizumab prescription in the Truven Medicaid claims during the identification period (07/07/2016 - 12/31/2018)
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — Omalizumab use was analyzed in two categories. First, initiators were defined as individuals with ≥ 1 omalizumab prescription. "Responders" were defined as individuals with at least 4 administrations of omalizumab.

SUMMARY:
A retrospective database pre-post cohort study, identifying asthmatic patients, aged 6- 11, with omalizumab use over 24 months

DETAILED DESCRIPTION:
This was a retrospective database pre-post cohort study, identifying asthmatic patients with omalizumab use over 24 months. Omalizumab use was analyzed in two categories. First, initiators were defined as individuals with ≥ 1 omalizumab claims. "Responders" were defined as individuals with at least 4 omalizumab claims. Descriptive statistics are provided for both groups, but outcomes are reported only for responders.

For this study, any persons from the Marketscan database with an asthma diagnosis and >= 1 omalizumab prescription/administration during the index period were identified. From this patient population the inclusion and exclusion criteria were applied, resulting in the final study cohort. Each person was assigned an index date based on their initial use of omalizumab.

Study Period: 07/07/2015 - 12/31/2019 Index Period: 07/07/2016 - 12/31/2018 Index Date: The date of the first medical or pharmacy claim of omalizumab Baseline Period (pre-index): 12 months before index date Follow up Period (post-index): 12 months after index date

The MarketScan® Claims Database (including commercial and Medicaid claims) was used. The claims database included data from 07/08/2015 - 12/31/2019. The MarketScan® Databases capture personspecific clinical utilization, expenditures, and enrollment across inpatient, outpatient, prescription drug, and carve-out services from a selection of large employers, health plans, and government and public organizations. The current study used the Commercial, Medicare Supplemental and Multi-State Medicaid Databases.

ELIGIBILITY:
Inclusion criteria:

We used all eligible Marketscan beneficiaries with an asthma diagnosis and omalizumab use between 07/07/2016 - 12/31/2018 (index period). Continuous enrollment in the Marketscan database was required to ensure the availability of claims data to capture study outcomes and covariates.

* Omalizumab cohort was defined as ≥1 prescription claims within the index period, with the date of first dispensing deemed the index date.
* Asthma was defined by ≥1 diagnosis code in any available diagnosis field on or prior to index date.

ICD-9-CM: 493.xx OR ICD-10-CM: J45.x

* 6-11 years of age at the time of index
* ≥12-months pre-index and ≥12-months post-index continuous eligibility in medical and pharmacy benefits
* Enrollment gap of ≤30 days will be considered continuous enrollment

Exclusion criteria:

Patients were excluded from the study if they had one or more of the following:

* Bronchial Thermoplasty at any time during data capture. Current Procedural Terminology (CPT): 31660, 31661
* Prior asthma-indicated biologic use during the 12 months pre or post-index

Omalizumab:

NDC: 50242004062; 50242004201 or HCPCS: J2357; S0107; C9217

Mepolizumab:

NDC: 00173088101, 00173088185 or HCPCS: J2182

Reslizumab:

NDC: 5931061031 or HCPCS: J2786

Benralizumab:

NDC: 0310173030 or HCPCS: C9466

Dupilumab:

NDC: 0024591400 or 0024591800

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: asthmatic patients, aged 6-11, with omalizumab use
Sampling Method: Probability Sample
Enrollment: 16246 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with uncontrolled asthma (impairment + risk criteria) post omalizumab treatment initiation | 12 months after index date (Index date defined as the date of the first medical or pharmacy claim of omalizumab between 07/07/2016 - 12/31/2018 index period)
  Uncontrolled asthma was based on either impairment or risk criteria in a 12- month consecutive period.
  * Impairment was identified as ≥6 Short-acting Beta Agonist (SABA) prescriptions dispensed in 12 months. Each prescription should reflect one month days supply.
  * Risk was defined as ≥1 unique exacerbation(s) in 12 months, including asthma-related ED visits or hospitalizations (emergency or hospital care with a diagnosis of asthma in the first position only [ICD-9 code 493.xx, ICD-10 code J45.xx]) or an OCS dispensing within 7 days AFTER an outpatient visit with an asthma diagnosis in ANY position.
  * The date of uncontrolled asthma assessment was defined as the earliest date between the sixth SABA prescription (impairment criteria) or the first exacerbation outcome during a consecutive 12-months (risk criteria).
Proportion of patients with excessive SABA use (≥6 SABA prescriptions dispensed in 12 months) (impairment criteria) | 12 months after index date (Index date defined as the date of the first medical or pharmacy claim of omalizumab between 07/07/2016 - 12/31/2018 index period)
  Proportion of patients with uncontrolled asthma (impairment criteria) were reported. Impairment was identified as ≥6 SABA prescriptions dispensed in 12 months. Each prescription should reflect one month days supply.
  - The date of uncontrolled asthma assessment was defined as the earliest date between the sixth SABA prescription (impairment criteria).
Proportion of patients with exacerbations requiring IP visits (risk criteria) | 12 months after index date (Index date defined as the date of the first medical or pharmacy claim of omalizumab between 07/07/2016 - 12/31/2018 index period)
  Proportion of patients with uncontrolled asthma (risk criteria) were reported. Risk was defined as ≥1 unique exacerbation(s) in 12 months, including asthma-related ED visits or hospitalizations (emergency or hospital care with a diagnosis of asthma in the first position only [ICD-9 code 493.xx, ICD-10 code J45.xx]) or an OCS dispensing within 7 days AFTER an outpatient visit with an asthma diagnosis in ANY position.
  - The date of uncontrolled asthma assessment was defined as the first exacerbation outcome during a consecutive 12-months (risk criteria).
Proportion of patients with exacerbations requiring ED visits (risk criteria) | 12 months after index date (Index date defined as the date of the first medical or pharmacy claim of omalizumab between 07/07/2016 - 12/31/2018 index period)
  Proportion of patients with uncontrolled asthma (risk criteria) were reported. Risk was defined as ≥1 unique exacerbation(s) in 12 months, including asthma-related ED visits or hospitalizations (emergency or hospital care with a diagnosis of asthma in the first position only [ICD-9 code 493.xx, ICD-10 code J45.xx]) or an OCS dispensing within 7 days AFTER an outpatient visit with an asthma diagnosis in ANY position.
  - The date of uncontrolled asthma assessment was defined as the first exacerbation outcome during a consecutive 12-months (risk criteria).
Proportion of patients with exacerbations requiring Oral corticosteroids (OCS) prescriptions (risk criteria) | 12 months after index date (Index date defined as the date of the first medical or pharmacy claim of omalizumab between 07/07/2016 - 12/31/2018 index period)
  Proportion of patients with uncontrolled asthma (risk criteria) were reported. Risk was defined as ≥1 unique exacerbation(s) in 12 months, including asthma-related ED visits or hospitalizations (emergency or hospital care with a diagnosis of asthma in the first position only [ICD-9 code 493.xx, ICD-10 code J45.xx]) or an OCS dispensing within 7 days AFTER an outpatient visit with an asthma diagnosis in ANY position.
  - The date of uncontrolled asthma assessment was defined as the first exacerbation outcome during a consecutive 12-months (risk criteria).
Mean daily dose of Inhaled Corticosteroids (ICS) use | 12 months after index date (Index date defined as the date of the first medical or pharmacy claim of omalizumab between 07/07/2016 - 12/31/2018 index period)
  Mean daily dose of Inhaled Corticosteroids (ICS) use was reported during the follow-up
Mean cumulative dose of OCS use | 12 months after index date (Index date defined as the date of the first medical or pharmacy claim of omalizumab between 07/07/2016 - 12/31/2018 index period)
  Mean cumulative dose of Oral corticosteroids were reported during follow-up
Mean number of prescriptions of OCS use | 12 months after index date (Index date defined as the date of the first medical or pharmacy claim of omalizumab between 07/07/2016 - 12/31/2018 index period)
  Mean number of prescriptions of OCS use were reported during follow-up
Mean days of supply of OCS use | 12 months after index date (Index date defined as the date of the first medical or pharmacy claim of omalizumab between 07/07/2016 - 12/31/2018 index period)
  Mean days of supply of OC were reported during follow-up

SECONDARY OUTCOMES:
Proportion of uncontrolled asthma patients (total: risk and impairment criteria) | through study completion, approximately 4 years (Study Period: 07/07/2015 - 12/31/2019)
  Uncontrolled asthma was based on either impairment or risk criteria in a 12- month consecutive period.
  * Impairment was identified as ≥6 Short-acting Beta Agonist (SABA) prescriptions dispensed in 12 months. Each prescription should reflect one month days supply.
  * Risk was defined as ≥1 unique exacerbation(s) in 12 months, including asthma-related ED visits or hospitalizations (emergency or hospital care with a diagnosis of asthma in the first position only [ICD-9 code 493.xx, ICD-10 code J45.xx]) or an OCS dispensing within 7 days AFTER an outpatient visit with an asthma diagnosis in ANY position.
  * The date of uncontrolled asthma assessment was defined as the earliest date between the sixth SABA prescription (impairment criteria) or the first exacerbation outcome during a consecutive 12-months (risk criteria).
Proportion of uncontrolled asthma patients (per impairment criteria) | through study completion, approximately 4 years (Study Period: 07/07/2015 - 12/31/2019)
  Proportion of patients with uncontrolled asthma (impairment criteria) were reported. Impairment was identified as ≥6 SABA prescriptions dispensed in 12 months. Each prescription should reflect one month days supply.
  - The date of uncontrolled asthma assessment was defined as the earliest date between the sixth SABA prescription (impairment criteria).
Proportion of uncontrolled asthma patients (per risk criteria) | through study completion, approximately 4 years (Study Period: 07/07/2015 - 12/31/2019)
  Risk was defined as ≥1 unique exacerbation(s) in 12 months, including asthma-related ED visits or hospitalizations (emergency or hospital care with a diagnosis of asthma in the first position only [ICD-9 code 493.xx, ICD-10 code J45.xx]) or an OCS dispensing within 7 days AFTER an outpatient visit with an asthma diagnosis in ANY position.
  - The date of uncontrolled asthma assessment was defined as the first exacerbation outcome during a consecutive 12-months (risk criteria).
Mean difference in the total number of asthma-related prescriptions | through study completion, approximately 4 years (Study Period: 07/07/2015 - 12/31/2019)
  Mean difference in the total number of asthma-related prescriptions between baseline and follow-up periods were reported
Mean difference in daily dose (of days supply) of ICS use | through study completion, approximately 4 years (Study Period: 07/07/2015 - 12/31/2019)
  Mean difference in daily dose (of days supply) between baseline and follow-up periods were reported
Proportion of patients with a reduction in daily dose of ICS use | through study completion, approximately 4 years (Study Period: 07/07/2015 - 12/31/2019)
  Proportion of patients with a reduction in daily dose between the baseline and follow-up periods were reported
Mean difference in daily dose of OCS use | through study completion, approximately 4 years (Study Period: 07/07/2015 - 12/31/2019)
  Mean difference in daily dose between baseline and follow-up periods were reported
Mean difference in number of prescriptions of OCS use | through study completion, approximately 4 years (Study Period: 07/07/2015 - 12/31/2019)
  Mean difference in number of prescriptions between baseline and follow-up periods were reported
Mean difference in days of supply of OCS use | through study completion, approximately 4 years (Study Period: 07/07/2015 - 12/31/2019)
  Mean difference in days of supply between baseline and follow-up periods were reported
Proportion of patients with a reduction in total prescriptions of OCS use | through study completion, approximately 4 years (Study Period: 07/07/2015 - 12/31/2019)
  Proportion of patients with a reduction in total prescriptions for OCS use between baseline and follow-up periods were reported

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigational Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CIGE025AUS55 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17888